CLINICAL TRIAL: NCT01475877
Title: Bromday (Bromfenac Ophthalmic Solution)0.09% QD vs Nevanac (Nepafenac Ophthalmic Suspension) 0.1% TID for Control of Pain and Epithelial Healing Post (PRK)
Brief Title: Bromday Versus Nevanac Eye Drops to Control Pain Following Photorefractive Keratectomy
Status: Completed | Type: Observational
Sponsor: Virdi Eye Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MAC-02-11
Record Dates: First submitted 2011-11-07; First posted 2011-11-21 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Myopia
Keywords: bromfenac; nepafenac; PRK; epithelial healing,
MeSH Terms: conditions — Myopia | interventions — bromfenac

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nepafenac
  Interventions: Drug: Bromfenac

INTERVENTIONS:
Drug: Bromfenac — Bromfenac 0.09% 1 drop in study eyes q day
  Other Names: Bromday

SUMMARY:
This study will compare the effect of two topical non-steroidal antiinflammatory agents to control pain after photorefractive keratectomy (PRK) eye surgery.

ELIGIBILITY:
Inclusion Criteria:

* male or female at least 18 years of age,
* no other ocular studies with 15 days prior to dosing,
* BCVA 20/200 or better,
* return for study visits and follow instructions from investigator and staff,
* self administer test article

Exclusion Criteria:

* Ocular inflammation,
* hypersensitivity to bromfenac or nepafenac,
* any corneal pathology,
* have had radial keratotomy,
* corneal transplant or corneal refractive surgery in the last two years

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing photorefractive keratectomy in both eyes
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Post-PRK pain | 7 days

SECONDARY OUTCOMES:
Post-PRK epithelial healing | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Navaneet S Borisuth, MD,PhD, Principal Investigator — Virdi Eye Clinic
Locations (1):
- Virdi Eye Clinic and Laser Vision Center, Rock Island, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
In the observational study conducted, there was no significant difference in pain levels or epithelial healing of post-photorefractive keratectomy patients who were treated with bromfenac 0.09% or nepafenac 0.1%